CLINICAL TRIAL: NCT01645228
Title: Could Non-invasive Biochemical, Image or Physiological Index Predict Significant Coronary Arterial Stenosis in Symptomatic Adults?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cathay General Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: CGH-P100133; NSC 101-2314-B-281 -007 (Other Grant/Funding Number: National Science Council, Taiwan)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- significant coronary artery stenosis: anyone coronary segment > 50% diameter stenosis
  Interventions: Radiation: coronary calcium score measurement; Biological: high sensitivity C reactive protein measurement; Procedure: ankle brachial index measurement

INTERVENTIONS:
Radiation: coronary calcium score measurement
Biological: high sensitivity C reactive protein measurement
Procedure: ankle brachial index measurement

SUMMARY:
To validate the capability of non-invasive bio-image tests in prediction of significant coronary stenosis of symptomatic adults.

DETAILED DESCRIPTION:
The main objective is to validate the capability of these non-invasive tests (CCS, hs-CRP and ABI) in prediction of significant coronary stenosis of symptomatic adults. The end-point will be the findings of coronary CT angiography. The investigators hope the results of our study could be applied on the interpretation of health examination and the advice of follow-up and therapy.

ELIGIBILITY:
Inclusion Criteria:

* subjects for a general health check-up protocol, which included CACS and CCTA, and biochemical measurements (total cholesterol, total triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, high sensitivity C reactive protein)

Exclusion Criteria:

* anyone allergy to iodine contrast medium, unable cooperation for CT scanning, asymptomatic

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: population for a general health check-up
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
coronary CT angiography | within one month

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Heng Mo, MD. PhD, Principal Investigator — Cathay General Hospital, Taiwan
Locations (1):
- Cathay General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Muntendam P, McCall C, Sanz J, Falk E, Fuster V; High-Risk Plaque Initiative. The BioImage Study: novel approaches to risk assessment in the primary prevention of atherosclerotic cardiovascular disease--study design and objectives. Am Heart J. 2010 Jul;160(1):49-57.e1. doi: 10.1016/j.ahj.2010.02.021. PMID 20598972
- [Background] Greenland P, Alpert JS, Beller GA, Benjamin EJ, Budoff MJ, Fayad ZA, Foster E, Hlatky MA, Hodgson JM, Kushner FG, Lauer MS, Shaw LJ, Smith SC Jr, Taylor AJ, Weintraub WS, Wenger NK, Jacobs AK, Smith SC Jr, Anderson JL, Albert N, Buller CE, Creager MA, Ettinger SM, Guyton RA, Halperin JL, Hochman JS, Kushner FG, Nishimura R, Ohman EM, Page RL, Stevenson WG, Tarkington LG, Yancy CW; American College of Cardiology Foundation; American Heart Association. 2010 ACCF/AHA guideline for assessment of cardiovascular risk in asymptomatic adults: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2010 Dec 14;56(25):e50-103. doi: 10.1016/j.jacc.2010.09.001. No abstract available. PMID 21144964
- [Background] Lim LS, Haq N, Mahmood S, Hoeksema L; ACPM Prevention Practice Committee; American College of Preventive Medicine. Atherosclerotic cardiovascular disease screening in adults: American College Of Preventive Medicine position statement on preventive practice. Am J Prev Med. 2011 Mar;40(3):381.e1-10. doi: 10.1016/j.amepre.2010.11.021. PMID 21335273
- [Background] Blaha MJ, Budoff MJ, DeFilippis AP, Blankstein R, Rivera JJ, Agatston A, O'Leary DH, Lima J, Blumenthal RS, Nasir K. Associations between C-reactive protein, coronary artery calcium, and cardiovascular events: implications for the JUPITER population from MESA, a population-based cohort study. Lancet. 2011 Aug 20;378(9792):684-92. doi: 10.1016/S0140-6736(11)60784-8. PMID 21856482
- [Background] Ridker PM. High-sensitivity C-reactive protein, vascular imaging, and vulnerable plaque: more evidence to support trials of antiinflammatory therapy for cardiovascular risk reduction. Circ Cardiovasc Imaging. 2011 May;4(3):195-7. doi: 10.1161/CIRCIMAGING.111.965053. No abstract available. PMID 21586741
- [Background] Murphy TP, Dhangana R, Pencina MJ, D'Agostino RB Sr. Ankle-brachial index and cardiovascular risk prediction: an analysis of 11,594 individuals with 10-year follow-up. Atherosclerosis. 2012 Jan;220(1):160-7. doi: 10.1016/j.atherosclerosis.2011.10.037. Epub 2011 Nov 3. PMID 22099055